CLINICAL TRIAL: NCT05866640
Title: A Prospective, Single-Arm, Single Center Feasibility Trial to Evaluate the Safety and Performance of the F2 Filter and Delivery System Used for Embolic Protection During Transcatheter Aortic Valve Replacement
Brief Title: Feasibility Trial of the F2 Filter and Delivery System for Embolic Protection During TAVR
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: EnCompass Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RG01
Record Dates: First submitted 2023-05-08; First posted 2023-05-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Aortic Stenosis
Keywords: TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Placement of the F2 device in the aorta to cover the great cerebral vessels.
  Interventions: Device: F2 filter and delivery system

INTERVENTIONS:
Device: F2 filter and delivery system — Placement of F2 device in aorta to cover great cerebral vessels

SUMMARY:
The goal of this clinical trial is to learn about the safety and performance of the F2 device for cerebral embolic protection in participants with symptomatic aortic stenosis underdoing a Transcatheter Aortic Valve replacement procedure.

Participants will complete several neurocognitive assessments and an MRI procedure.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the safety and performance of the F2 device for cerebral embolic protection in participants with symptomatic aortic stenosis underdoing a transcatheter aortic valve replacement procedure. The F2 device is inserted via a transfemoral approach and positioned in the aorta to cover and protect the three great cerebral vessels from any debris released during the valve replacement procedure. The F2 device remains in place during the aortic valve replacement procedure. After the valve is placed, the F2 device is removed.

ELIGIBILITY:
Inclusion Criteria:

criteria:

1. Age ≥ 22 years.
2. The patient meets the established criteria and indications for commercially available TAVR (Edwards/Medtronic) for transfemoral access.
3. Montreal Cognitive Assessment (MoCA) score ≥ 26 at screening.
4. The patient is willing and able to comply with protocol-specified follow-up evaluations.
5. The patient or legally authorized representative is able and willing to provide written informed consent.

Exclusion Criteria:

1. Contraindications to MRI (e.g., subjects with MR unsafe implants including implantable temporary or permanent pacemaker or defibrillator, metal implants in field of view, metallic fragments, clips, or devices in the brain or eye before TAVR procedure, or claustrophobia).
2. Severe peripheral arterial, abdominal aortic, or thoracic aortic disease that precludes delivery sheath vascular access or filter deployment.
3. Patients in whom the aortic arch is heavily calcified, severely atheromatous, or severely tortuous.
4. Ascending aortic diameter > 38 mm or transverse aortic diameter > 27 mm.
5. Evidence of an acute myocardial infarction within 1 month before TAVR.
6. Pre-existing prosthetic heart valve or prosthetic ring in any position.
7. Known intracardiac thrombus.
8. Severe allergy or known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel, nitinol, stainless steel alloy, and/or contrast sensitivity that cannot be adequately pre-medicated.
9. History of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated.
10. Patients who refuse blood transfusion.
11. Active peptic ulcer or history of upper gastrointestinal (GI) bleeding within the prior 3 months.
12. Recent (within 6 months) CVA or a TIA.
13. Renal insufficiency (creatinine > 2.5 mg/dL or GFR < 30) and/or renal replacement therapy at the time of screening.
14. Patients with hepatic failure (Child-Pugh class C).
15. Patients with hypercoagulable states that cannot be corrected by additional periprocedural heparin.
16. Patients presenting with cardiogenic shock or requiring vasopressor or inotropic support at the time of the index procedure.
17. Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20%.
18. Life expectancy < 12 months.
19. Currently participating in an investigational drug or another device study that has not completed the initial primary endpoint evaluation (e.g., long term follow-up study/continued access study subjects are able to be included).
20. Subjects who have had treatment with any other investigational device within 30 days prior to study enrollment.
21. Planned surgery or invasive procedure within 30 days following the index procedure (TAVR with F2 Filter).
22. Patients planned to undergo any other cardiac surgical or interventional procedure (e.g., concurrent coronary revascularization) during the TAVR procedure or within 10 days prior to the TAVR procedure. NOTE: Balloon valvuloplasty during TAVR is permitted. Diagnostic cardiac catheterization is permitted within 10 days prior to the TAVR procedure.
23. Patients with known mental or physical illness or known history of substance abuse that may cause non-compliance with the protocol or confound the data interpretation.
24. Females who are pregnant or nursing or plan to become pregnant during their participation in the study. Female subjects of child-bearing potential must have a negative pregnancy test at screening.
25. Any other condition that in the opinion of the investigator, precludes study participation or poses a significant hazard to the patient.

    -

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | 30 days
  Major adverse cardiac and cerebrovascular events

SECONDARY OUTCOMES:
New lesions | 8-72 hours
  total new lesion volume, average individual new lesion volume, number of new lesions, location of new lesions, territory of new lesions
Performance | intra-procedure
  technical success (% of patients with successful device deployment, position and retreival and procedure success (% of patients with technical device success and no device-related safety events)
Modified Rankin Scale | 30 day
  Measures neurological disability on scale of 0-6 (low score is better outcome)
National Institute of Health Stroke Scale | 30 day
  Measures stroke severity on scale of 0 - 42 (low score is better outcome)
Montreal Cognitive Assessment | 30 day
  Measures cognitive impairment on scale of 0 - 30 (high score is better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Duhay, MD, Study Director — Sponsor GmbH
Locations (1):
- Healthycore, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No